CLINICAL TRIAL: NCT04512235
Title: A Phase 3, Double-Blind, Multicenter Study to Evaluate the Efficacy and Safety of CAEL-101 and Plasma Cell Dyscrasia Treatment Versus Placebo and Plasma Cell Dyscrasia Treatment in Plasma Cell Dyscrasia Treatment Naïve Patients With Mayo Stage IIIa AL Amyloidosis
Brief Title: A Study to Evaluate the Efficacy and Safety of CAEL-101 in Patients With Mayo Stage IIIa AL Amyloidosis (CARES)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAEL101-302
Record Dates: First submitted 2020-08-10; First posted 2020-08-13 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: AL Amyloidosis
Keywords: Plasma Cell Dyscrasia; cyclophosphamide, bortezomib and dexamethasone (CyBorD); AL Amyloidosis; Amyloid, Light chain Amyloidosis; treatment-naïve; Mayo Stage IIIa
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis; Paraproteinemias | interventions — Cyclophosphamide; Bortezomib; Dexamethasone; Clinical Protocols

STUDY DESIGN:
Intervention Model Description: This is a double-blind, randomized, multicenter, international Phase 3 study of CAEL-101 combined with SoC PCD treatment versus placebo combined with SoC PCD treatment in Mayo stage IIIa PCD treatment-naïve AL amyloidosis patients. Approximately 267 patients will be enrolled using a 2:1 randomization ratio and stratification will be based on geographic region across investigator sites. The primary evaluation treatment period (PETP) part of the study will stop when the last patient is randomized in the PETP plus 18 months. Patients in both study intervention groups will be followed from randomization until death from any cause, heart transplant, left valve assist device (LVAD) implantation or until end of study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blind, randomized, multicenter international Phase 3 study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CAEL-101 combined with SoC plasma cell dyscrasia (Experimental): The study is divided into 2 parts, the Primary Study and the Open-Label Extension Study. CAEL-101 is administered as an intravenous (IV) infusion over approximately 2 hours. It is planned that all patients will continue their double-blind treatment until the last patient is randomized in the study plus 18 months.
  Interventions: Drug: CAEL-101; Drug: cyclophosphamide, bortezomib, and dexamethasone (CyBorD) regimen
- Placebo combined with SoC plasma cell dyscrasia (Placebo Comparator): Patients randomized to receive placebo will receive 0.9% normal saline in an equivalent volume to a CAEL-101 infusion (approximately 250 cc). It is planned that all patients will continue their double-blind treatment until the last patient is randomized in the study plus 18 months.
  Interventions: Other: Placebo; Drug: cyclophosphamide, bortezomib, and dexamethasone (CyBorD) regimen

INTERVENTIONS:
Drug: CAEL-101 — The investigational product, CAEL-101, is formulated as a sterile liquid solution of protein plus excipients for dilution in a single-use, stoppered, glass vial. Each 10 mL vial contains 300 mg of CAEL-101 at a concentration of 30 mg/mL. CAEL-101 will be diluted with commercially available 0.9% Normal Saline.
  Other Names: Anselamimab
  Arms: CAEL-101 combined with SoC plasma cell dyscrasia
Other: Placebo — Commercially available 0.9% Normal Saline will be used as the placebo.
  Arms: Placebo combined with SoC plasma cell dyscrasia
Drug: cyclophosphamide, bortezomib, and dexamethasone (CyBorD) regimen — According to institutional standard of care.
  Other Names: Anselamimab

SUMMARY:
AL (or light chain) amyloidosis begins in the bone marrow where abnormal proteins misfold and create free light chains that cannot be broken down. These free light chains bind together to form amyloid fibrils that build up in the extracellular space of organs, affecting the kidneys, heart, liver, spleen, nervous system and digestive tract.

The primary purpose of this study is to determine whether CAEL-101, a monoclonal antibody that removes AL amyloid deposits from tissues and organs, improves overall survival, reduces cardiovascular related hospitalizations and it is safe and well tolerated in patients with stage IIIa AL amyloidosis.

DETAILED DESCRIPTION:
This is a double-blind, randomized, multicenter international Phase 3 study of CAEL-101 combined with standard of care (SoC) plasma cell dyscrasia (PCD) treatment versus placebo combined with SoC PCD treatment in Mayo stage IIIa PCD treatment-naïve AL amyloidosis patients. Approximately 267 patients will be enrolled using a 2:1 randomization ratio. Patients in both study intervention groups will be followed from randomization until death from any cause, heart transplant, left valve assist device (LVAD) implantation or until the end of study.

ELIGIBILITY:
Key Inclusion Criteria:

* AL amyloidosis stage IIIa based on the European Modification of the 2004 Standard Mayo Clinic Staging who also have NT-proBNP > 650 ng/L at the time of Screening
* Measurable hematologic disease at Screening as defined by at least one of the following:

  1. Involved/uninvolved free light chain difference (dFLC) > 4 mg/dL or
  2. Involved free light chain (iFLC) > 4 mg/dL with abnormal Kappa/Lambda ratio or
  3. Serum protein electrophoresis (SPEP) m-spike > 0.5 g/dL
* Histopathological diagnosis of amyloidosis based on polarizing light microscopy of green bi-refringent material in Congo red stained tissue specimens AND confirmation of AL derived amyloid deposits by at least one of the following:

  1. Immunohistochemistry/Immunofluroescence
  2. Mass spectrometry or
  3. Characteristic electron microscopy appearance/Immunoelectron microscopy
* Cardiac involvement as defined by:

  a. Documented clinical signs and symptoms supportive of a diagnosis of heart failure in the setting of a confirmed diagnosis of AL amyloidosis in the absence of an alternative explanation for heart failure AND b. At least one of the following: i. Endomyocardial biopsy demonstrating AL cardiac amyloidosis or ii. Echocardiogram demonstrating a mean left ventricular wall thickness (calculated as [IVSd+LPWd]/2) of > 12 mm at diastole in the absence of other causes (e.g., severe hypertension, aortic stenosis), which would adequately explain the degree of wall thickening or iii. Cardiac magnetic resonance imaging (MRI) with gadolinium contrast agent diagnostic of cardiac amyloidosis
* Planned first-line treatment for plasma cell dyscrasia is a cyclophosphamide-bortezomib-dexamethasone (CyBorD)-based regimen administered as SoC
* Women of childbearing potential (WOCBP) must have a negative pregnancy test during Screening and must agree to use highly effective contraception from Screening to at least 5 months following the last study drug administration or 12 months following the last dose of her PCD therapy, whichever is longer
* Men must be surgically sterile or must agree to use highly effective contraception from Screening to at least 5 months following the last study drug administration or 12 months following the last dose of his PCD therapy, whichever is longer

Key Exclusion Criteria:

* Have any other form of amyloidosis other than AL amyloidosis
* Received prior therapy for AL amyloidosis or multiple myeloma. A maximum exposure of 2 weeks of a CyBorD-based PCD treatment after Screening laboratory samples are obtained and prior to randomization is allowed.
* Has POEMS (plasma cell dyscrasia with polyneuropathy, organomegaly, endocrinopathy, monoclonal protein and skin changes) syndrome or multiple myeloma defined as clonal bone marrow plasma cells > 10% from a bone marrow biopsy (performed ≤ 3 months prior to signing the ICF) or biopsy-proven (performed ≤ 3 months prior to signing the ICF) bony or extramedullary plasmacytoma AND one or more of the following CRAB features:

  a. Evidence of end organ damage that can be attributed to the underlying plasma cell proliferative disorder (eg, multiple myeloma and POEMS syndrome) specifically: i. Hypercalcemia: serum calcium > 0.25 mmol/L (> 1 mg/dL) higher than the upper limit of normal (ULN) or > 2.75 mmol/L (> 11 mg/dL) OR ii. Renal insufficiency: creatinine clearance < 40 mL per minute or serum creatinine > 177 umol/L (> 2 mg/dL) OR iii. Anemia: hemoglobin value of > 20 g/L below the lowest limit of normal, or a hemoglobin value < 100 g/L OR iv. Bone lesions: one or more osteolytic lesion on imaging tests (performed ≤ 3 months prior to signing the ICF): skeletal radiography, computed tomography (CT), or positron emission tomography (PET)/CT, or MRI. If bone marrow has < 10% clonal plasma cells, more than one bone lesion is required to distinguish from solitary plasmacytoma with minimal marrow involvement OR b. Any one of the following biomarkers of malignancy: i. 60% or greater clonal plasma cells on bone marrow examination OR ii. More than one focal lesion on MRI that is at least 5 mm or greater in size
* Have supine systolic blood pressure < 90 mmHg or symptomatic orthostatic hypotension, defined as a decrease in systolic blood pressure upon standing of > 30 mmHg despite medical management (e.g., midodrine, fludrocortisones) in the absence of volume depletion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 284 (Actual)
Dates: Start 2020-11-03 (Actual); Primary Completion 2025-04-08 (Actual); Study Completion 2027-04-08 (Estimated)

PRIMARY OUTCOMES:
A hierarchical combination of Time to All-cause Mortality and Frequency of Cardiovascular hospitalizations | From the date of randomization to date of death or Primary Evaluation Treatment Period (PETP) (up to 54 months)
Number of Participants with Treatment emergent Adverse Events (TEAEs) | From date of randomization to Primary Evaluation Treatment Period (PETP) (up to 59 months)

SECONDARY OUTCOMES:
Time to All-cause Mortality | From the date of randomization to date of death or Primary Evaluation Treatment Period (PETP) (up to 54 months)
Frequency of cardiovascular-related hospitalizations (CVH) | From the date of randomization to date of death or Primary Evaluation Treatment Period (PETP) (up to 54 months)
Change From Baseline to Week 50 in the Kansas City Cardiomyopathy Questionnaire-Overall Score (KCCQ-OS) | Baseline, Week 50
  A 23-item self-administered questionnaire that quantifies physical function, symptoms, social function, self-efficacy and knowledge and quality of life. It requires an average of 4-6 minutes to complete and uses an ordinal, adjectival (Likert) scale. Patients will provide their level of agreement or disagreement with a agree-disagree scale for a series of statements. This questionnaire captures how the patients feel physically. Scores range from 0 to 100, where higher scores reflected better health status (fewer symptoms, fewer social or physical limitations, and better quality of life)
Change from Baseline to Week 50 in N-Terminal Pro-B-type Natriuretic Peptide (NT-proBNP) in blood samples | Baseline, Week 50
  To assess improvement in cardiomyopathy as measured by NT-proBNP. For each participant, blood sample will be assayed for NT-proBNP, comparing the participant's baseline value over time to assess improvement in the heart by reduced amyloidosis as measured by an increase or decrease in amyloidosis-related biomarkers: NT-proBNP.
Change From Baseline to Week 50 in Global Longitudinal Strain (GLS%) | Baseline, Week 50
  To assess improvement in heart function as measured by percent Global Longitudinal Strain (GLS%). GLS% is a non-invasive imaging technique to assess heart function where a higher/lower percentage is indicative of improvement.
Change From Baseline to Week 50 in Distance Walked (in Meters) during a Six-minute Walk Test (6MWT) | Baseline, Week 50
  The 6MWT measures the distance a patient can quickly walk on a flat, hard surface in a period of 6 minutes. It evaluates the global and integrated response of all the systems involved during exercise. This is a self-paced test; patients choose their own intensity of exercise and are allowed to stop and rest during the test.
Change From Baseline to Week 50 in the Short Form-36 (SF-36) Version 2 (v2) Physical Component Score (PCS) | Baseline, Week 50
  A self-administered questionnaire containing 36 items that measures health on functional status, well-being and overall evaluation of health in 8 domains. It requires approximately 5 minutes to complete and uses scaled, ordinal responses (e.g., All of the time, Most of the time, A good bit of the time, etc.).

CONTACTS AND LOCATIONS:
Overall Officials: Scott Swenson, MD, Study Director — Alexion, AstraZeneca Rare Disease
Locations (102):
- United States (29):
  - Research Site, Scottsdale, Arizona
  - Research Site, Duarte, California
  - Research Site, Palo Alto, California
  - Research Site, San Francisco, California
  - Research Site, Jacksonville, Florida
  - Research Site, Weston, Florida
  - Research Site, Indianapolis, Indiana
  - Research Site, New Orleans, Louisiana
  - Research Site, Baltimore, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, Rochester, Minnesota
  - Research Site, St Louis, Missouri
  - Research Site, New York, New York
  - Research Site, Rochester, New York
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Durham, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Cleveland, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Nashville, Tennessee
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Seattle, Washington
  - Research Site, Madison, Wisconsin
  - Research Site, Milwaukee, Wisconsin
- Australia (4):
  - Research Site, Box Hill
  - Research Site, Murdoch
  - Research Site, Westmead
  - Research Site, Woolloongabba
- Austria (2):
  - Research Site, Linz
  - Research Site, Vienna
- Belgium (2):
  - Research Site, Anderlecht
  - Research Site, Leuven
- Brazil (3):
  - Research Site, Porto Alegre
  - Research Site, Ribeirão Preto
  - Research Site, Salvador
- Canada (2):
  - Research Site, Calgary, Alberta
  - Research Site, Toronto, Ontario
- China (7):
  - Research Site, Beijing
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Shanghai
  - Research Site, Suzhou
  - Research Site, Wenzhou
  - Research Site, Wuhan
- Czechia (2):
  - Research Site, Ostrava Poruba
  - Research Site, Prague
- France (13):
  - Research Site, Caen
  - Research Site, Créteil
  - Research Site, Dijon
  - Research Site, Lille
  - Research Site, Limoges
  - Research Site, Marseille
  - Research Site, Paris
  - Research Site, Pessac
  - Research Site, Pierre-Bénite
  - Research Site, Poitiers
  - Research Site, Rennes
  - Research Site, Toulouse
  - Research Site, Tours
- Germany (6):
  - Research Site, Berlin
  - Research Site, Düsseldorf
  - Research Site, Essen
  - Research Site, Hamburg
  - Research Site, Heidelberg
  - Research Site, Würzburg
- Greece (3):
  - Research Site, Athens
  - Research Site, Rio
  - Research Site, Thessaloniki
- Israel (5):
  - Research Site, Haifa
  - Research Site, Jerusalem
  - Research Site, Petah Tikva
  - Research Site, Tel Aviv
  - Research Site, Tel Litwinsky
- Research Site, Brescia, Italy
- Japan (8):
  - Research Site, Fukushima
  - Research Site, Kanazawa
  - Research Site, Kashiwa-shi
  - Research Site, Kita-ku
  - Research Site, Kumamoto
  - Research Site, Matsumoto-shi
  - Research Site, Nagoya
  - Research Site, Shibuya-ku
- Poland (2):
  - Research Site, Gdansk
  - Research Site, Warsaw
- Research Site, Saint Petersburg, Russia
- Research Site, Seoul, South Korea
- Spain (9):
  - Research Site, Barcelona
  - Research Site, Gijón
  - Research Site, Granada
  - Research Site, Madrid
  - Research Site, Majadahonda
  - Research Site, Pamplona
  - Research Site, Salamanca
  - Research Site, Seville
  - Research Site, Valencia
- United Kingdom (2):
  - Research Site, Glasgow
  - Research Site, London

IPD SHARING:
Plan to Share IPD: Yes
Each patient will be assigned a unique identifier after signing the Informed Consent Form (ICF). Patient numbers will not be reassigned. Any patient records or datasets transferred to the Sponsor must contain only the unique identifier and must not include patient names or any information which would make the patient identifiable. Patients will be informed that their personal study-related data will be used by the Sponsor in accordance with local data protection laws and that their medical records may be examined by representatives of the Sponsor, Institutional Review Board (IRB)/Independent Ethics Committee (IEC) members and by inspectors from regulatory authorities. Study monitors will inspect all documents and records that are required to be maintained by the Investigator for this study.